CLINICAL TRIAL: NCT03571009
Title: Utilization of Real-time Pain Monitoring System (PAMS), ANAPA System, in Patients With Rheumatic Disease
Brief Title: Real-time Pain Monitoring in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ji Hyeon Ju (Other)
Responsible Party: Sponsor-Investigator, Ji Hyeon Ju, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PAAS in FMS
Record Dates: First submitted 2018-06-04; First posted 2018-06-27 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Pain; Fibromyalgia
MeSH Terms: conditions — Pain; Fibromyalgia

STUDY DESIGN:
Intervention Model Description: The patients were supposed to complete three visits (baseline, one month, and three months). Patients in the PAAS group were provided with a wearable device (Painmeter, LST, Seoul, Korea) and smartphone application (DrKooB-PAAS, iKooB Inc. Seoul, South Korea), while the control group was provided conventional treatment without using the system. After screening, patients were randomly assigned to a group with an opaque envelope that contained the written randomization result. After completing the three months of the study, patients in the control group were then allocated to the PAAS group and underwent three additional months of study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- utilization of PAAS (Experimental): conventional treatment utilization of PAAS
  Interventions: Device: utilization of PAAS
- Conventional care (No Intervention): conventional treatment only

INTERVENTIONS:
Device: utilization of PAAS — utilization of real-time pain assessment and analysis system (PAAS) consists of wearing device and reporting a real-time pain using the device
  Arms: utilization of PAAS

SUMMARY:
This study aims to examine whether the pain of fibromyalgia patients can be reduced with utilization of real-time pain monitoring system (PAAS). In this pilot study, adult fibromyalgia patients were randomly assigned to use or to not use PAAS. Changes in the visual analogue scale (VAS) were examined by rheumatologists at baseline and after three months, and correlations between conventional pain VAS or PAAS VAS and clinical parameters (patient global assessment, physician global assessment, fibromyalgia impact questionnaire) were investigated. We also examined if the utilization of PAAS can affect health related quality of life and depression.

DETAILED DESCRIPTION:
Chronic pain is difficult to treat and is debilitating to patients in various ways, including wide spread suffering, disability, social displacement, and expense. For effective pain management, the first step should be to assess the exact status of the pain. This process may include characterizing the pain, quantifying it as accurately as possible, and analyzing influencing factors. However, it is hard to objectify pain because it is an invisible and subjective. The visual analogue scale (VAS) is widely used to assess the severity of pain. Moreover, current management of chronic pain is based on a patient's recall, which may be inaccurate. It would be ideal if we could manage pain by recording its status on a real-time basis, reflecting the impact of environmental factors. The Pain Assessment and Analysis System (PAAS) has been developed to monitor and record real-time pain. Users are asked to report the type of experienced pain and its severity. Therefore, for user convenience, PAAS can be accessed using a wearable device (Painmeter, LST, Seoul, Korea) that is interlinked with a smartphone mobile application (DrKooB-PAAS, iKooB Inc. Seoul, South Korea). The system records the frequency and severity of pain and can create reports summarizing the pain over the course of various time intervals. In addition, this system also records the time, temperature, humidity, and weather, along with the reported pain, to determine any correlations between the pain and these environmental factors. Fibromyalgia (FMS) is a complex disorder characterized by intractable, widespread pain and somatic symptoms such as insomnia, constipation, diarrhea, and cognitive dysfunction. The exact pathogenesis has yet to be elucidated, but current understandings suggest that disturbances in pain-regulating neurotransmitters are involved. The diagnosis and management of FMS are a challenge for physicians. Its management should combine pharmacological and non-pharmacological approaches, which suggests there are various factors that influence treatment outcomes. To date, tricyclic agents, serotonin norepinephrine reuptake inhibitors, and pregabalin are known to have beneficial effects; however, a substantial number of patients are still suffering from the uncontrolled pain of FMS.

To address the pain in these patients, an appropriate pain monitoring system that can reflect real-time pain severity and frequency and can analyze the pattern of impacting factors can be used to provide effective treatment and to eventually improve patient pain. Therefore, we aimed to investigate the feasibility of a real-time pain monitoring system, the Pain Assessment and Analysis System (PAAS), in patients with FMS in order to evaluate its effect on pain reduction. In addition, we evaluated the correlations between the VAS measured by PAAS and clinical parameters reflecting the disease activity of FMS.

ELIGIBILITY:
* Inclusion Criteria:

  19 years of age or older diagnosed with fibromyalgia based on the 2010 American College of Rheumatology preliminary diagnostic criteria for FMS
* Exclusion Criteria:

previously diagnosed with a serious systemic medical illness a medical condition that can affect bodily pain: eg. (1) inflammatory arthritis (2) malignancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Changes in Pain visual analogue scale | 3 months after randomization
  The pain visual analogue scale (0-10 mm) of the patient is addressed on each visit. Changes in pain visual analogue scale on 3 months visit is evaluated.

SECONDARY OUTCOMES:
Changes in the dose of medication | 3 months after baseline visit
  To address the dose and the class of the medication
Changes in the disease activity | 3 months after baseline visit
  Fibromyalgia impact questionnaire is used to address the disease activity
Changes in the quality of life | 3 months after baseline visit
  Euro QoL - 5D questionnaire is used to address hearth related quality of life
Changes in the depressive symptoms | 3 months after baseline visit
  Beck's depression index is used to address the severity of depressive symptoms
Correlation of pain visual analogue scale (VAS) by pain assessment analysis system (PAAS) with patient global assessment | 1 month after baseline visit
  correlation between PAAS VAS and patient global assessment (0-10 mm)
Correlation of pain visual analogue scale (VAS) by pain assessment analysis system (PAAS) with disease activity | 1 month after baseline visit
  correlation between PAAS VAS and Fibromyalgia impact questionnaire scores
Correlation of pain visual analogue scale (VAS) by pain assessment analysis system (PAAS) with physician global assessment | 1 month after baseline visit
  correlation between PAAS VAS and physician global assessment (0-10 mm)

CONTACTS AND LOCATIONS:
Overall Officials: Ji Hyeon Ju, MD PhD, Principal Investigator — Seoul St. Mary's Hospital

IPD SHARING:
Plan to Share IPD: Undecided